CLINICAL TRIAL: NCT00406302
Title: Multicenter Phase II Study Evaluating Docetaxel, CDDP, and Cetuximab as Induction Regimen Prior to Surgery in Chemo-naive Patients With NSCLC Stage IB, II and IIIA
Brief Title: Immune Response on Neoadjuvant Therapy in Non-small-cell Lung Cancer (NSCLC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Wolfgang Hilbe (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); Sanofi (Industry); TAKO - Tiroler Arbeitskreis Onkologie (Unknown)
Responsible Party: Sponsor-Investigator, Wolfgang Hilbe, Ao. Univ. Prof. Dr., Medical University of Vienna
Organization: Medical University of Vienna (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2006-004639-31
Record Dates: First submitted 2006-12-01; First posted 2006-12-04 (Estimated); Last update posted 2014-04-29 (Estimated); Status verified 2014-04

CONDITIONS: Carcinoma, Non-small-cell Lung
Keywords: NSCLC; non-small-cell lung cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Docetaxel; Oxaliplatin; Cetuximab; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Docetaxel — 75mg/m², day 1,22
  Other Names: Taxotere
Drug: oxaliplatin — 40mg/m², d1,2,22,23
  Other Names: CDDP
Drug: cetuximab — 400mg/m² (day1), 250mg/m² (day 8,15,22,29,36)
  Other Names: Erbitux
Procedure: surgery — 28 days after end of induction chemotherapy

SUMMARY:
Primary objective is to assess the overall response rate (ORR) after induction therapy with docetaxel in combination with CDDP and cetuximab in patients with NSCLC stage IB, II, and IIIa. ORR will be determined by the percentage of patients achieving objective response rates (CR + PR) according to the RECIST guidelines.

DETAILED DESCRIPTION:
Primary objective is to assess the overall response rate (ORR) after induction therapy with docetaxel in combination with CDDP and cetuximab in patients with NSCLC stage IB, II, and IIIa. ORR will be determined by the percentage of patients achieving objective response rates (CR + PR) according to the RECIST guidelines.

Secondary objective is

* To evaluate pathological response determined by histological work up of the surgical specimens according to TNM stages.
* To evaluate the metabolic response determined by PET analysis.
* To assess overall survival (OS) (median survival time and percentage of 1-year survival). OS is defined as time elapsed from the date of patient inclusion until recorded date of death.
* To characterize and quantify toxic effects of the scheduled therapy. Safety profile and tolerability will be assessed by recording adverse events, clinically significant laboratory abnormalities, physical examination and vital signs. Toxicities will be evaluated according to the NCI-CTC Toxicity Criteria and adverse events which are not reported in NCI-CTC will be graded as mild, moderate, severe or life-threatening. All patients who received any of the scheduled therapy will be included in the overall toxicity analysis.
* To evaluate the immunological response determined by regulatory T-cells and immune activation markers, to define chemoresistance by pharmacogenomic testing.

ELIGIBILITY:
Inclusion Criteria:

Histology and staging of the disease

* Histological confirmed NSCLC; histology may include: large cell, squamous cell or adenocarcinoma but no SCLC.
* Anatomically and functionally resectable NSCLC stage IB (T2N0) stage II (T1-2 N1, T3 N0) or stage IIIA (T3 N1) (see TAKO guidelines 2006, www.tako.or.at)
* Measurable disease according to RECIST criteria

General conditions

* 18-80 years.
* WHO 0-2; life expectancy of more than 3 months
* Effective contraception for both male and female patients if the risk of conception exists
* Adequate respiratory function, sufficient for necessary surgical treatment
* Adequate hematological function (Hb > 10 g/dl, ANC > 2.0 x 10 9/L, platelets > 100 x 10 9/L).
* Adequate renal and hepatic functions: total bilirubin within normal limits, serum creatinine within normal limits, in case of limit value the creatinine clearance should be > 60 ml/min, ASAT and ALAT < 2.5 x UNL, alkaline phosphatase < 5 x UNL.

Initial work-up

* Complete initial work-up within three weeks prior to first infusion includes chest CT scan, abdominal CT-scan, brain CT scan if indicated, PET-scan, bronchoscopy and mediastinoscopy, pulmonary function. Within 7 days prior to inclusion laboratory investigations and biological work up.
* Signed initial consent prior to protocol specific procedures.

Exclusion Criteria:

Diagnosis

* Evidence of brain metastases or other distant metastasis equivalent to stage IV disease
* History of prior malignancies, except for curatively treated non-melanoma skin cancer or in situ carcinoma of the cervix or other curatively treated cancer with no evidence of disease for at least five years
* Other serious concomitant illness or medical condition:
* Congestive heart failure or angina pectoris, except if medically controlled, history of myocardial infarction within 1 year from study entry, uncontrolled hypertension or arrhythmia
* History of significant neurological or psychiatric disorders, including dementia or seizure
* Active infection requiring i.v. antibiotics
* Active ulcer, unstable diabetes mellitus or other contraindications to corticotherapy
* Current peripheral neuropathy WHO grade > 2

Prior or concurrent therapy

* Prior chemotherapy or immunotherapy for NSCLC
* Prior surgery or radiotherapy for NSCLC
* Concurrent treatment with other experimental drugs, unapproved medical procedures or other anticancer therapy
* Concurrent continuous treatment with systemic steroids for antiemetic use, intermittent application is allowed

General conditions

* Pregnant (absence to be confirmed by ß-HCG-test) or lactating patients
* Patients (M/F) with reproductive potential not implementing adequate contraceptive measurements
* Participation in other clinical trials with experimental agents or non approved medical procedures during study and within 30 days prior to study entry
* Psychological, familial, sociological or geographical conditions which do not permit medical follow-up and compliance with the study protocol.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2007-01; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
overall response rate (complete plus partial response) according to RECIST guidelines | June 2011

SECONDARY OUTCOMES:
Pathological response | June 2011
Metabolic response | June 2011
Immunological response | June 2011
Overall survival | June 2011
Safety profile and tolerability | June 2011
overall response rate (complete plus partial response) according to RECIST guidelines | June 2011

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang Hilbe, Prof. Dr., Principal Investigator — University Hospital Innsbruck, Internal Medicine
Locations (7):
- Austria (7):
  - University Hospital, Internal Medicine, Innsbruck, Tyrol
  - Hosptial Kufstein, Kufstein, Tyrol
  - Hospital Natters, Natters, Tyrol
  - Hospital Zams, Zams, Tyrol
  - Prim. Dr. Bolitschek, Linz
  - Prim. Dr. H. Schinko, Linz
  - OA Dr. Rainer Kolb, Wels

REFERENCES:
- [Background] Fossella F, Pereira JR, von Pawel J, Pluzanska A, Gorbounova V, Kaukel E, Mattson KV, Ramlau R, Szczesna A, Fidias P, Millward M, Belani CP. Randomized, multinational, phase III study of docetaxel plus platinum combinations versus vinorelbine plus cisplatin for advanced non-small-cell lung cancer: the TAX 326 study group. J Clin Oncol. 2003 Aug 15;21(16):3016-24. doi: 10.1200/JCO.2003.12.046. Epub 2003 Jul 1. PMID 12837811
- [Background] Rosell R., et al. Proc Am Soc Clin Oncol 23: 618, 2004
- [Background] Betticher DC, et al. Proc Am Soc Clin Oncol: 1824, 1999